CLINICAL TRIAL: NCT02343796
Title: Clinical Follow-up of Direct/Indirect Bridge, Orthodontic and Periodontal Splint Applications by Using Fibre-reinforced Composite.
Brief Title: Clinical Follow-up of Direct/Indirect Bridge, Orthodontic and Periodontal Splint by Using Fibre-reinforced Composite
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Ovul Kumbuloglu, Associate Professor, Ege University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-9.1/4
Record Dates: First submitted 2015-01-07; First posted 2015-01-22 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Tooth Loss; Tooth Mobility
Keywords: Fiberglass reinforced resins
MeSH Terms: conditions — Tooth Loss; Tooth Mobility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fibre-reinforced composite (Experimental): Fibreglass reinforced composite restoration-everStick as a medical device intervention will be applied on each subject by using either direct or indirect method. everStick (GC, Belgium) will be used as a fibre reinforcement material.
  Interventions: Other: Fibreglass reinforced composite restoration-everStick; Device: everStick

INTERVENTIONS:
Other: Fibreglass reinforced composite restoration-everStick — For those subjects with space availability on interocclusal distance, composite resin restorations with fibreglass reinforcement will be applied without any tooth preparation by using adhesive techniques.
Device: everStick — GC, Belgium

SUMMARY:
The purpose of this study is to determine whether fibre-reinforced composite resin restorations are effective for single tooth replacement, elimination of tooth mobility following periodontal treatment and as an orthodontic retainer.

DETAILED DESCRIPTION:
Adhesive dentistry is based on preventive dental approach. In presence of such advanced and minimally invasive techniques, destructive treatment methods should not be preferred for clinical situations, such as missing single tooth cases, tooth mobility following periodontal treatment and prevention of relapse after orthodontic treatments. Glass fibre is a reinforcement material, and increases the flexibility of the material together which it has been used. Fibre-reinforced applications by using direct or indirect techniques. This material and method is easily applicable, biocompatible, repairable and economical on a high extent.

ELIGIBILITY:
Inclusion Criteria:

* referring patients for missing tooth replacement or fixation of tooth mobility following periodontal treatment or maintenance of teeth in corrected positions following orthodontic treatment

Exclusion Criteria:

* insufficient interocclusal distance
* poor oral hygiene

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2003-06; Primary Completion 2014-12 (Actual); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with clinical survival of the applied restoration, splint or retainer, as indicated by observations for any fractures on composite. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Ovul Kumbuloglu, Assoc Prof, Principal Investigator — Ege University
Locations (1):
- Ege University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
IPD would be considered for sharing with other reseachers during manuscript preparation.

REFERENCES:
- [Background] Kumbuloglu O, Ozcan M, User A. Fracture strength of direct surface-retained fixed partial dentures: effect of fiber reinforcement versus the use of particulate filler composites only. Dent Mater J. 2008 Mar;27(2):195-202. doi: 10.4012/dmj.27.195. PMID 18540392